CLINICAL TRIAL: NCT06112977
Title: Restore-B: A Mixed-methods Trial Evaluating the Feasibility of a Multi-centre Randomised Controlled Trial Comparing No-mesh to Mesh-assisted Immediate Prepectoral Implant-based Breast Reconstruction
Brief Title: Restore-B: A Trial Comparing Prepectoral Implant-based Breast Reconstruction With and Without Mesh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Restore-B
Record Dates: First submitted 2023-10-10; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer; Risk Reduction
Keywords: Breast surgery; Breast Reconstruction; Prepectoral; Implant; Mesh; Acellular dermal matrix
MeSH Terms: conditions — Breast Neoplasms; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Restore-B is a prospective, multicentre parallel 2-armed single-blinded randomised controlled feasibility trial comparing no-mesh to mesh- assisted immediate implant-based prepectoral breast reconstruction surgery.
  Patients will be randomised 1:1 to either the intervention surgery (no- mesh) arm or the control arm surgery (mesh-assisted).
Who Masked: Participant
Masking Description: Participants will be blinded to their surgical allocation (mesh or no mesh) and will be unblinded after completion of their post-operative questionnaire at day 90.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate prepectoral implant-based breast reconstruction without surgical mesh. (Active Comparator): Prepectoral implant (expander or fixed volume) breast reconstruction without mesh
  Interventions: Procedure: Prepectoral implant-based immediate breast reconstruction
- Immediate prepectoral implant- based breast reconstruction with surgical mesh (Active Comparator): Prepectoral implant (expander or fixed volume) breast reconstruction with mesh (biological or synthetic)
  Interventions: Procedure: Prepectoral implant-based immediate breast reconstruction

INTERVENTIONS:
Procedure: Prepectoral implant-based immediate breast reconstruction — Prepectoral implant based breast reconstruction is an immediate breast reconstruction whereby a fixed volume implant or expander is placed on top of the chest wall muscle (Pectoralis Major) to reconstruct the breast after mastectomy.

SUMMARY:
The goal of this feasibility randomised controlled clinical trial (RCT) is to compare mesh-assisted to no-mesh pre-pectoral implant based immediate breast reconstruction in women undergoing mastectomy for treatment of breast cancer or for risk reduction of an inherited breast cancer risk.

The main questions it aims to answer are:

* To determine the feasibility of a definitive RCT comparing the clinical and cost- effectiveness of no- mesh versus mesh- assisted pre-pectoral breast reconstruction.
* To determine if it is possible to collect data to inform a future economic analysis on the use of mesh in breast reconstruction.

Participants will be randomly allocated to have their breast reconstruction either with the use of mesh or without the use of mesh prior to the start of the operation. Participants will be blinded to their allocation until day 90 post operatively. Participants will be asked to have medical photography and to complete a short quality of life questionnaire before and after surgery at 90 days prior to finding out their allocation.

DETAILED DESCRIPTION:
Trial Design:

Restore-B is a prospective, multicentre parallel 2-armed single-blinded randomised controlled feasibility trial comparing no-mesh to mesh- assisted immediate implant-based prepectoral breast reconstruction surgery.

Patients will be randomised 1:1 to either the intervention surgery (no- mesh) arm or the control arm surgery (mesh-assisted).

Planned Trial Period:

The overall period of the trial is:

12 months recruitment, 3 months follow-up and 6 months data analysis and final reporting of results.

Trial Participants:

Women over 18 years old eligible for elective immediate prepectoral implant-based breast reconstruction with mesh for cancer treatment or risk reduction surgery

Intervention:

Immediate prepectoral implant-based (implant or expander) breast reconstruction without surgical mesh (ADM or synthetic).

Comparator:

Immediate prepectoral implant- based (implant or expander) breast reconstruction with surgical mesh (ADM or synthetic) (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years
* Participant is able and willing to give informed consent for participation in the trial
* Eligible for immediate prepectoral implant-based breast reconstruction with implant or expander with mesh (biologic or synthetic) for cancer treatment or risk reduction surgery.
* In the Investigator's opinion, can comply with all trial requirements.

Exclusion Criteria:

The participant may not enter the trial if any of the following apply:

* Participant is pregnant, lactating or planning pregnancy during the trial
* Patient refusal
* Delayed breast reconstruction post simple mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a definitive RCT comparing the clinical and cost- effectiveness of no- mesh versus mesh- assisted pre-pectoral breast reconstruction. | 16 months
  * Number of patients eligible
  * Number of patients consented and randomised within 12 months recruitment
  * Number of patients lost to follow up/withdrawal
  * Completeness of data per participant (%)

SECONDARY OUTCOMES:
Clinical outcomes in each arm | 90 days
  - Number of clinical complications in each arm up to 90 days: seroma, infection, re-operation, haematoma, mesh removal, implant removal, revision surgery
Patient reported outcome: Breast-Q Breast Reconstruction Quality of Life (QoL) Measure | 90 days post operatively
  Breast Q measures health related QoL and patient satisfaction in the context of breast surgery. The breast reconstruction module will be used in this study and measured pre- and post-operatively in each arm.
  All BREAST-Q scales are transformed into scores that range from 0-100, independent of the type and number of modules. The scores are computed by adding the response items together and then converting the raw sum scale score to a score from 0-100. For all BREAST-Q scales, a higher score means greater satisfaction or better QOL (depending on the scale).
Patient reported outcome: EuroQoL-EQ5D Quality of Life (QoL) Measure | 90days post operatively
  Quality of life (QoL) questionnaires pre-and post-operatively at 90 days measured by EuroQol-EQ5D-5L.
  This QoL questionnaire comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems (1-5). The patient is asked to indicate her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A higher score indicates more severe or frequent problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ms Rachel Rolph, MBBS MA FRCS, Principal Investigator — University of Oxford
Locations (1):
- Surigcal Intervention Trials Unit (SITU), Nuffield Department of Surgical Sciences, University of Oxford, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published for reference. Study outcome data will be published at the end of the trial. Data will determine progression to full RCT.
Supporting Information: Study Protocol
Time Frame: 3 months. Available long term
Access Criteria: Open access publication of the protocol in British Medical Journal Open Scientific Journal.

REFERENCES:
- [Derived] Rolph R, Ziebland S, Cook JA, Iglesias C, Wakefield-Scurr J, Malyon C, Scaife J, Taylor A, Hennessy A, Markham S, Bernstein M, Douek M; Restore-B Feasibility Collaborative Group. Prepectoral no mesh versus mesh immediate implant-based reconstruction after mastectomy (Restore-B): a multicentre single-blinded randomised controlled feasibility study protocol. BMJ Open. 2025 Oct 17;15(10):e103278. doi: 10.1136/bmjopen-2025-103278. PMID 41106857